CLINICAL TRIAL: NCT01514019
Title: An Open-label, Single-dose, Two-treatment, Randomized, Cross-over Study to Investigate the Effects of the SLCO2B1 c.1457C>T Polymorphism and Apple Juice on the Pharmacokinetics and Pharmacodynamics of Acebutolol in Healthy Korean and Japanese Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: In-Jin Jang, MD, PhD (Other)
Collaborators: Oita University (Other); Seoul National University Hospital (Other); Kyushu University (Other)
Responsible Party: Sponsor-Investigator, In-Jin Jang, MD, PhD, Professor of Clinical Pharmacology and Therapeutics, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2012_Acebutolol
Record Dates: First submitted 2012-01-17; First posted 2012-01-20 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Healthy
Keywords: SLCO2B1 genotype; effect of apple juice
MeSH Terms: interventions — Acebutolol; Lactose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acebutolol (Experimental): Acebutolol 200 mg capsule (Acetanol®)
  Interventions: Drug: Acebutolol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acebutolol — Acebutolol
  Other Names: Acebutolol 200 mg capsule (Acetanol®)
  Arms: Acebutolol
Drug: Placebo — Placebo capsule(Capsules filled up with lactose)
  Other Names: Placebo capsule(Capsules filled up with lactose)
  Arms: Placebo

SUMMARY:
An open-label, single-dose, two-treatment, randomized, cross-over study to investigate the effects of the SLCO2B1 c.1457C>T polymorphism and apple juice on the pharmacokinetics and pharmacodynamics of acebutolol in healthy Korean and Japanese volunteers

ELIGIBILITY:
Inclusion Criteria:

* Subject is informed of the investigational nature of this study and voluntarily agrees to participate in this study and signs an Institutional Review Board (IRB) - approved informed consent prior to performing any of the screening procedures

Exclusion Criteria:

* A subject with history of allergies including study drug (acebutolol) or other drug allergies (aspirin, antibiotics, etc.), or history of clinically significant allergies

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
AUC of acebutolol according to the SLCO2B1 genotypes | 0-24 hr after drug administration
  The area under the plasma concentration versus time curve, from time 0 to the last measurable concentration, as calculated by the linear/log trapezoidal method will be summarized by treatment and genotype group using descriptive statistics.

SECONDARY OUTCOMES:
Blood pressure of the subjects who administered acebutolol according to the SLCO2B1 genotypes | 0-24 hr after drug admnistration
  Blood pressure (systolic, diastolic) measurement will be presented as descriptive statistics for the difference from baseline where appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Kyoichi Ohashi, MD, PhD, Study Chair — Department of Clinical Pharmacology and Therapeutics, Oita University Faculty of Medicine, Oita, Japan
Locations (2):
- General Clinical Research Center, Oita University Hospital, Ōita, Japan
- Seoul National University Hospital, Seoul, South Korea